CLINICAL TRIAL: NCT00375947
Title: Efficacy of a Home-Based Hand Range-of-Motion and Strength Training Exercise Program for Improvement of Hand Function in Older Adults With Hand Osteoarthritis: a Randomized Controlled Trial
Brief Title: Study of Effectiveness of Hand Exercises to Treat Symptoms of Hand Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Arthritis Research Institute of America (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ARIA-0001
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Osteoarthritis
Keywords: exercise; hand disability; arthritis; AUSCAN
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Arthritis

ARMS (2):
- 1 (Experimental): Home-based hand exercise program
  Interventions: Other: Hand Exercise
- 2 (Placebo Comparator): Sham hand cream
  Interventions: Other: sham hand cream

INTERVENTIONS:
Other: Hand Exercise
  Arms: 1
Other: sham hand cream — placebo intervention
  Arms: 2

SUMMARY:
Participants in this study will do hand exercises once per day for 16 weeks. The purpose of the study is to determine if hand exercises designed to improve range of movement and strength are an effective way to decrease functional limitations for people with hand osteoarthritis. The study will also attempt to determine if pain and stiffness are improved, and if hand strength and dexterity are improved.

DETAILED DESCRIPTION:
Osteoarthritis is one of the most common joint disorders in the elderly, yet few studies have targeted symptomatic osteoarthritis, especially symptomatic hand osteoarthritis.

Hand OA is a chronic disease for which no cure is currently available, the symptomatic pharmacologic treatment has significant side effects , and none of the recommended passive modality physical therapies have been demonstrated to improve function. To this end, our study constitutes a systematic approach to show how patients with hand OA might benefit from an intervention that is free of side effects, easily administered, and readily acceptable.

STUDY OBJECTIVE: To evaluate the efficacy of exercise for the reduction of hand functional disability associated with hand osteoarthritis that is both symptomatic and radiographic.

Intervention activity: A 16-week, home-based exercise program designed to decrease physical impairment of the hands. The exercise routine consists of nine (9) exercises performed once daily, bilaterally. The program will take about 10-20 minutes to complete. Six (6) exercises involve active range-of-motion (AROM) and three (3) involve hand and finger flexion using a Thera-Band ® Hand Exerciser (Hygenic Corporation, Akron, OH). The Hand Exerciser is a polymer ball with resistance that varies by color, with yellow 'extra soft' at approximately 1.5 lbs when 50% compressed, red "soft" at 3 lbs, green "medium" at 5 lbs, and blue "firm" at 8 lbs. The Hand Exerciser comes in two sizes; "regular" will be used for small to average sized hands and "extra large" for larger hands. The starting resistance for each subject will be determined by baseline grip and pinch static strength testing. Those with weaker grip or key pinch will use a softer ball, stronger subjects will use medium or firm, per predetermined standards. Some subjects may use more than one color of ball depending on clinical presentation (e.g., greater pain and dysfunction in MCP may require softer ball for pinching exercises, while a firmer ball is appropriate for gripping). A study booklet with written instructions and photos will describe how to perform the exercises.

Control activity: Application of a fragrance-free non-therapeutic topical cream, applied once daily. A study booklet with written instructions and photos will describe how to apply the cream.

Order of activities in this crossover study is assigned randomly using a random number table.

There will be a 16-week washout period of no intervention between the two treatment periods, regardless of the order in which the subjects began using the treatments. The washout period is designed to allow all measures to return to original baseline as much as possible.

The study will be 48 weeks in duration (three 16-week periods). Subjects will be enrolled as a dynamic entry cohort. Subjects are to note any adverse reactions to the exercises or the topical hand cream. They are to report such to the principal investigator of the trial. All subjects will be asked to complete a Participation Log. This will give study investigators a surrogate measure of participation and compliance.

As well as collecting information concerning demographics, medications, and relevant medical and social history at baseline, at each assessment participants will be asked to complete the AUSCAN Index (Australian Canadian Osteoarthritis Hand Index (AUSCAN) [Bellamy, 2002]). The AUSCAN Index is a self-administered questionnaire that assesses the three dimensions of pain, joint stiffness, and disability due to hand osteoarthritis using a battery of 15 questions. Scaled on 5-point Likert scales and 100mm Visual Analog Scales, the AUSCAN 3.1 is a valid, reliable and responsive measure of outcome. The index has been subject to validation studies that have addressed the following clinometric issues: reliability - stability, internal consistency; validity - face, content, construct; and responsiveness. The 100mm VA Scale will be used in the current study.

At baseline and 16 weeks of each of the two treatment periods (exercise and and cream) subjects' maximum grip, key pinch, and 3-point pinch strengths will be assessed using Jamar® grip and pinch dynamometers (Sammons Preston Rolyan, Bolingbrook, IL). Dexterity will be measured using standard tests of the Purdue Peg Board (Lafayette Instruments, Lafayette, IN).

Data collection schedule

The AUCSAN Index will be administered after a subject has completed specified lengths of participation. All participants will be assessed three times during both the exercise and hand cream intervention periods.

1. Baseline
2. 8 weeks
3. 16 weeks

In addition, bilateral hand grip, key pinch, & 3-point pinch maximum strength, and hand dexterity (all best of 3 trials) will be tested at two points during each of the two intervention periods.

1. Baseline
2. 16 weeks

STATISTICAL METHODS

Statistical analysis will be performed using SAS statistical software (version 9.12, Cary, NC). Group differences of change between baseline and 16 weeks in hand function will be compared. Values and scores will be tested for Gaussian distribution (normality test). If the data are normally distributed, a parametric test (paired t-test) will be used. If the data are not normally distributed, a non-parametric test (signed ranks test) will be used. Data will be analyzed per intent-to-treat.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Ages 50 years and older
* Reside within Tampa Bay Region, Florida
* Presence of symptomatic OA as determined by the AUSCAN Index. Specifically, a hand function score of > 225 mm for the AUSCAN VA-subscale
* Presence of radiographic hand OA, as defined by grades 2, or higher, per the Kellgren and Lawrence scale in one or more joints.

Exclusion Criteria:

* Concomitant rheumatic disease (e.g., rheumatoid arthritis, gout, lupus, fibromyalgia)
* Current hand or wrist injury (e.g., carpal tunnel syndrome, palmer tenosynovitis, fracture, sprain)
* Use of an assistive device such as a cane or crutch
* Has hand surgery scheduled within the 48 weeks following the start of the study
* Prior hand surgery requiring joint replacement or other instrumentation in the hands
* Received any intra-articular injection (hyaluronic acid, corticosteroid, or joint lavage) during the 3 months preceding the study
* Currently participating in another conflicting research study
* Currently using a therapeutic hand cream or practicing a hand exercise routine
* Unwilling to sign an informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2005-11; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Australian-Canadian Osteoarthritis Index (AUSCAN)hand disability score at 16 weeks of exercise

SECONDARY OUTCOMES:
AUSCAN hand pain score at 16 weeks of exercise
AUSCAN hand stiffness score at 16 weeks of exercise
Maximal and average grip strength at 16 weeks of exercise
Maximal and average key pinch strength at 16 weeks of exercise
Maximal and average 3-point pinch strength at 16 weeks of exercise
Purdue Peg Board dexterity scores at 16 weeks of exercise

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Rogers, MS, Principal Investigator — The Arthritis Research Institute of America; Frances V Wilder, PhD, Study Director — The Arthritis Research Institute of America
Locations (1):
- The Arthritis Research Institute of America, Clearwater, Florida, United States

REFERENCES:
- See also: ARIA web site — http://www.preventarthritis.org